CLINICAL TRIAL: NCT01608516
Title: Multimodal Assessment of the Inflammatory Atheromatous Plaque : Comparison Between 68Ga-NODAGA-RGD PET/CT, 18F-FDG PET/CT, MRI AND US
Brief Title: Multimodal Imaging Assessment of the Inflammatory Atheromatous Plaque
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Principal Investigator, John O. Prior, Chief of Department of Nuclear Medicine, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 80/10
Record Dates: First submitted 2012-04-16; First posted 2012-05-31 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Inflammation; Atheromatous Plaques; Carotid Artery Diseases
Keywords: PET/CT; 68Ga-NODAGA-RGD; 18F-FDG; MRI; US ultrasound; inflammatory atheromatous plaque; endarterectomy
MeSH Terms: conditions — Inflammation; Plaque, Atherosclerotic; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NODAGA-RGD radiotracer (Experimental): All patients will undergo a 68Ga-NODAGA-RGD PET/CT, a 18F-FDG PET/CT, a MRI and a US.
  Interventions: Drug: 68Ga-NODAGA-RGD PET/CT

INTERVENTIONS:
Drug: 68Ga-NODAGA-RGD PET/CT — 200 MBq 68 Ga-NODAGA-RGD will be administered i.v. and images centred on the carotid area acquired

SUMMARY:
The present study aims at assessing the ability of 68Ga-NODAGA-RGD PET/CT for the detection of inflammatory atheromatous plaques in the carotid arteries, compared to 18F-FDG PET/CT, MRI and US and to determine the contribution of each imaging technique. Current gold standard for inflammation is histopathology.

Hypothesis : 68Ga-NODAGA-RGD might give a better initial evaluation of patients with atheromatous plaques in the carotid artery eligible for endarterectomy.

DETAILED DESCRIPTION:
Patients with indication for endarterectomy will be presented the present protocol. If inclusion criteria are fulfilled, patients will have a 18F-FDG PET/CT + carotid US performed 6 to 2 days before endarterectomy and 68Ga-NODAGA-RGD PET/CT + MRI performed the day before endarterectomy. Histopathological sample will be analyzed to measure plaque inflammation.

All imaging results and histopathology results will be pooled and compared.

ELIGIBILITY:
Inclusion Criteria:

* age <= 85 years
* Karnofsky >= 80%
* patient with indication ofr carotid endarterectomy
* signed consent form

Exclusion Criteria:

* indication for surgery other than endarterectomy <14 days
* contraindication to surgery
* contraindication to MRI
* contraindication to gadolinium injection (stage 4/5 kidney insufficiency, GFR<30ml/min/1.73m2)
* pregnancy, breastfeeding
* lack of discernment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of each method of imaging for the detection of inflammatory atheromatous plaques | Within1 month of endarterectomy
  The potential of each of the methods of imaging for the detection of inflammatory atheromatous plaques will be compared. For that purpose, the capacity of every criterion of primary assessment to determine the presence of an unstable plaque will be studied compared with the histopathological sample.

SECONDARY OUTCOMES:
Comparison of AUC of the imaging methods | Within1 month of endarterectomy
  A comparison of the AUC will be realized to determine the superiority of a method compared with the other one, by a non parametric test comparing AUC , ROC curves respectively.
Analysis of histopathological sample of endarterectomy | Within1 month of endarterectomy
  The histopathological analysis will be the degree of local inflammation estimated by the macrophagic infiltration as well as the degree of neovascularization.

CONTACTS AND LOCATIONS:
Overall Officials: John O. Prior, PhD, MD, Principal Investigator — Lausanne University Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gnesin S, Mitsakis P, Cicone F, Deshayes E, Dunet V, Gallino AF, Kosinski M, Baechler S, Buchegger F, Viertl D, Prior JO. First in-human radiation dosimetry of 68Ga-NODAGA-RGDyK. EJNMMI Res. 2017 Dec;7(1):43. doi: 10.1186/s13550-017-0288-x. Epub 2017 May 18. PMID 28523582